CLINICAL TRIAL: NCT05048654
Title: A Novel Ovarian Reserve Monitoring Algorithm for Patients at Risk of Ovarian Injury From Gonadotoxic Therapy
Acronym: MA
Status: Withdrawn | Type: Observational
Why Stopped: Cancelled by PI
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 21-3085
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Diseases; Fertility Issues; Gonadal Disorders
MeSH Terms: conditions — Ovarian Diseases; Infertility; Gonadal Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: Retrospective: Retrospectively, there will be an abstract of AMH and FSH from survivors seen at CHCO and UCH from October 1st, 2016 to September 31st, 2019 and assess time points.
- Group B: Prospective: Prospectively, survivors will be evaluated by a member of the FPRLE team in the outpatient clinic at 12 months post-therapy completion and every 6 months to 36 months as part of clinical care. Per standard of care AMH and FSH will be drawn at each time point.

SUMMARY:
This is an observational cohort study to examine the use of a novel proposed ovarian reserve monitoring algorithm to (1) identify patients who are at risk of DOR and POI from gonadotoxic therapy, (2) minimize time from treatment to utilization of assisted reproductive technologies, and (3) improves prognosis for successful ART based on AFC for patients who pursue fertility or fertility preservation.

DETAILED DESCRIPTION:
Study Design: This is an observational cohort study to examine the use of a novel proposed ovarian reserve monitoring algorithm to (1) identify patients who are at risk of DOR and POI from gonadotoxic therapy, (2) minimize time from treatment to utilization of assisted reproductive technologies, and (3) improves prognosis for successful ART based on AFC for patients who pursue fertility or fertility preservation.

Group B: Prospectively, survivors will be evaluated by a member of the FPRLE team in the outpatient clinic at 12 months post-therapy completion and every 6 months to 36 months as part of clinical care. AMH and FSH will be drawn at each time point.

Group A: Retrospectively, we will abstract AMH and FSH from survivors seen at CHCO and UCH from October 1st, 2016 to September 31st, 2019 and assess time points.

Approach Aim 1: The Investigator will assess AMH and FSH in both groups and evaluate whether the monitoring algorithm allows for early identification of DOR prior to the occurrence of POI. The investigator will calculate time from end of treatment to diagnosis of DOR and POI to evaluate if the monitoring algorithm detects these conditions earlier than historical controls.

Statistical analysis: The investigator will provide descriptive statistics and time to event analysis by group.

Aim 2: The Investigator will assess time from end of treatment to utilization of ART as defined by ovulation induction with or without insemination, in vitro fertilization, and/or third-party reproduction.

Statistical analysis: The Investigator will provide descriptive statistics and time to event analysis by group (A and B).

Aim 3: The Investigator will assess if early identification of DOR improves prognosis for successful ART for Group B as compared to Group A. The Investigator define success as an AFC greater than or equal to 6 at time of evaluation by REI.

Statistical analysis: The Investigator will provide descriptive statistics for the prevalence of AFC greater than 6 by group (A and B).

Aim 4: The Investigator will characterize barriers to utilization of ART by surveying participants who were referred to REI. The Investigator will assess the following: (1) if participants declined or accepted referral, (2) if they accepted, were they successful, and (3) if they declined, reasons for declining.

ELIGIBILITY:
Inclusion Criteria:

* · Female patients ages 8 - 39 years of age

  * Seen in CHCO or AMC outpatient clinics for any of the following reasons:

    * At risk for fertility problems (Z91.89)
    * Encounter for fertility preservation counseling (Z31.62)
    * Primary ovarian insufficiency
    * Premature ovarian failure/premature menopause
    * Diminished ovarian reserve
  * At least 12 months post-completion of chemotherapy and/or radiation
  * History of a fertility-threatening diagnosis receiving chemotherapy; radiation; or surgery to the reproductive organs for malignancy, including but not limited to:

    * Any type of cancer/malignancy
    * Rheumatoid arthritis
    * Systemic lupus erythematosus
    * Aplastic anemia
    * Fanconi anemia
    * Diamond-Blackfan syndrome
    * Hurler syndrome
    * Other autoimmune conditions

Exclusion Criteria:

* Disorders of sexual development (i.e., gonadal dysgenesis, Turner syndrome/mosaicism, etc.)
* History of bilateral oophorectomy
* Transgender patients not receiving chemotherapy; radiation; or surgery to the reproductive organs for malignancy
* Inability to consent/assent

Ages: 8 Years to 39 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes — This study address female population as it is looking at Ovarian reserves only
Study Population: Study participants will be pre- and post-pubertal females 8 years and older greater seen at the University of Colorado Anschutz Pavilion and/or Children's Hospital Colorado who have received gonadotoxic chemotherapy; radiation; or surgical excision of a reproductive organ for malignancy. The anticipated study population for Group B will be approximately 3,338 per year for five years for an projected total of 16, 690. Group A will have an anticipated study population of 3,338 per year for three years for an projected total of 10,014. For Groups A and B that is a grand total of 26,704.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Does the novel monitoring algorithm (intervention group) detect early Ovarian disfunction | 2 year follow up
  We will compare ovarian reserve categories (normal, diminished ovarian reserve, primary ovarian insufficiency), defined using AMH and FSH, in a retrospective group using the standard of care and a prospective group using a new monitoring algorithm.

SECONDARY OUTCOMES:
Time to ART | 2 year follow up
  Assess if the length of time from end of treatment to utilization of ART is different between the two groups.
Evaluate if there is an improved AFC in the new monitoring algorithm group | 2 year follow up
  Assess if the proportion of AFC greater than or equal to 6 at time of evaluation by REI is higher in the new monitoring algorithm group compared to the standard of care.
Characterizing barriers to utilization of ART | 2 year year follow up
  We will examine the following: (1) if participants declined or accepted referral, (2) if they accepted, were they successful, and (3) if they declined, reasons for declining.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Appiah, MD, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No